CLINICAL TRIAL: NCT04725279
Title: Usefulness of Rehabilitation in Patients With Cervical Imbalance. Use of Stabilometric Platform and Motion Sensors. (Provisional Title)
Brief Title: Usefulness of Rehabilitation in Patients With Cervical Imbalance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Marco Polo Royo, Principal Investigator, Universidad de Zaragoza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MPolo
Record Dates: First submitted 2021-01-17; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Rehabilitation; Cervical Vertigo
MeSH Terms: interventions — Electric Stimulation Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Type of rehabilitation treatment (Experimental): Depending on whether the cervical pain associated with vertigo in the patients associated pain radiating to the arms or not, treatment with conventional physiotherapy or electrotherapy was prescribed. In addition, both groups had a control group that performed exercises at home prescribed by a physician.
  Interventions: Procedure: Rehabilitation Treatment: Physiotherapy, Electrotherapy or Exercises at home

INTERVENTIONS:
Procedure: Rehabilitation Treatment: Physiotherapy, Electrotherapy or Exercises at home — The 67 patients attended the rehabilitation consultation where, after taking the anamnesis, they began to perform balance tests with a stabilometric platform and those patients with associated neck pain, with cervical motion sensors. Treatment with conventional physiotherapy, electrotherapy or exercises at home was prescribed as appropriate to each one. 3 months later, the patients were examined again in consultation, using a new anamnesis, the platform and the sensors.

SUMMARY:
Using the data obtained in a study carried out at the Hospital of Alcañiz (Teruel, Spain) between February and July 2019, with a stabilometric platform and with movement sensors, the investigators want to demonstrate that the rehabilitation works in those patients with vertigo or dizziness of cervical origin. For this, the data obtained from that sample, which was of 67 patients, will be analyzed in a pre-post rehabilitation treatment study, objectifying whether the patients improved or not, both in terms of imbalance and cervical pain, if any.

DETAILED DESCRIPTION:
Using the data obtained in a study carried out at the Hospital of Alcañiz (Teruel, Spain) between February and July 2019, with a stabilometric platform and with movement sensors, the investigators want to demonstrate that the rehabilitation works in those patients with vertigo or dizziness of cervical origin. For this, the data obtained from that sample, which was of 67 patients, will be analyzed in a pre-post rehabilitation treatment study, objectifying whether the patients improved or not, both in terms of imbalance and cervical pain, if any. The 67 patients attended the rehabilitation consultation where, after taking the anamnesis, they began to perform balance tests with a stabilometric platform and those patients with associated neck pain, with cervical motion sensors. Treatment with conventional physiotherapy, electrotherapy or exercises at home was prescribed as appropriate to each one. 3 months later, the patients were examined again in consultation, using a new anamnesis, the platform and the sensors. With the data obtained in said field work, carried out in 2019, the present study aims to analyze the usefulness of rehabilitation treatment in vertigo.

ELIGIBILITY:
Inclusion Criteria:

* Present vertigo of vestibular, neurological or cervical cause.
* The last episode of vertigo occurred less than a year ago.

Exclusion Criteria:

* Present acute musculoskeletal pathology in the lower limbs or lumbar spine.
* Present some lower limb amputation.
* Present unresolved visual pathology.
* Being active with anticancer treatment.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Number of patients who improve, worsen or do not present changes after rehabilitation treatment | 3 months passed between the first evaluation and the second.
  It is evaluated whether the patients, after undergoing the corresponding prescribed rehabilitation treatment, are better, worse or the same as before undergoing it.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Ciencias de la Salud, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No
Data from the 67 patients who were part of the study will not be shared with anyone who did not participate in the study.